CLINICAL TRIAL: NCT01369654
Title: Development and Pilot Test of an Elective Bilateral Salpingo-Oophorectomy (BSO) Decision Support Guide
Acronym: BSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 10-03107
Record Dates: First submitted 2011-06-06; First posted 2011-06-09 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Surgical Procedure, Unspecified
Keywords: hysterectomy with Bilateral Salpingo Oophorectomy; Oophorectomy; Gynecologic condition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computerized decision aid (Experimental)
  Interventions: Behavioral: Computerized decision aid with 1 type of value clarification

INTERVENTIONS:
Behavioral: Computerized decision aid with 1 type of value clarification — Women will be instructed to view a computerized BSO decision support guide.
  Other Names: Computerized decision aid with 2 types

SUMMARY:
The investigators propose to conduct formative research to gain an understanding of patients' needs and desires regarding elective Bilateral Salpingo-Oophorectomy (BSO) decision making, and to develop and pilot test a BSO Decision Support Guide, in preparation for a randomized, controlled trial of the effect of this decision aid on decision quality and use of BSO. The proposed study will consist of 3 phases. In phase 1, the investigators plan to conduct focus groups among women who have had a hysterectomy with or without bilateral salpingo-oophorectomy (BSO) to gain an understanding of what they understood about BSO and its possible outcomes at the time of their hysterectomy and what they would have liked to have known, the extent and manner in which they were included in decision making regarding BSO, and how they feel about the decision now. The investigators also will collect qualitative data from women who are scheduled for hysterectomy and currently facing the decision whether or not to undergo elective BSO. In phase 2, the investigators plan to create a BSO Decision Support Guide using information obtained from the literature, from our formative research, and the experience of providers who have counseled women about this choice. In phase 3, the investigators plan to pilot test the BSO Decision Support Guide among women scheduled to undergo hysterectomy for benign conditions to assess its usefulness and usability for patients and their providers and to prepare for a randomized study of its impact on decision quality and use of BSO. 62 women who are scheduled to undergo hysterectomy for a non-cancerous uterine condition will participate in the pilot study. These women will participate in a baseline interview, during which they will be provided access to the BSO Decision Support Guide, and 2 follow up telephone interviews (one as they are making their final BSO decision and a second after they have undergone and recovered from their hysterectomy (with or without BSO). Data will be used to generate the final version of the Decision Support Guide, to finalize evaluation measures for future studies of the effectiveness of the guide, and to determine effect sizes for the outcomes of knowledge, BSO use, decision satisfaction and decisional conflict.

DETAILED DESCRIPTION:
Specific Aim 1) Conduct formative research to assess how sociodemographically diverse women who will be undergoing hysterectomy for non-cancerous conditions view elective BSO and to assess their information needs and desires regarding shared decision making in this context.

Specific Aim 2) Create a BSO Decision Support Guide using information obtained from the literature, from our formative research, and the experience of providers who have counseled women about this choice.

Specific Aim 3) Pilot test the BSO Decision Support Guide among women scheduled to undergo hysterectomy for benign conditions to assess its usefulness and usability for patients and their providers and to prepare for a randomized study of its impact on decision quality and use of BSO.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal defined as having at least one menses in the 3 months prior to surgery;
* age >40 years;
* Plans to undergo an elective hysterectomy for symptomatic fibroids, abnormal bleeding, pelvic pain, or pelvic organ prolapse;
* Plans to undergo hysterectomy via any route (laparoscopic, laparotomy, or vaginal;
* speaks English

Exclusion Criteria:

* having personal or family history of breast and/or ovarian cancer or a known breast cancer gene (BRCA) mutation;
* Known or suspected adnexal mass by exam or radiologic imaging;
* Gynecologist recommends BSO for treatment of pelvic pain and/or endometriosis;
* Diagnosis of coronary heart disease (CHD) or osteoporosis;
* Cannot speak English;
* Less than 40 years of age.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Satisfaction with Intervention | 6 months
  After study participants participate in a baseline interview, during which they will be provided access to the BSO Decision Support guide, they will receive 2 follow up telephone interviews (one as they are making their final BSO decision and a second after they have undergone and recovered from their hysterectomy (with or without BSO)

SECONDARY OUTCOMES:
BSO Decisional conflict, regret, anxiety | 6 months
  In the 2nd follow up telephone interview we will ask how helpful was the BSO Decision Support Guide, and if they have any conflicts or regrets with the decisions made.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Kuppermann, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States